CLINICAL TRIAL: NCT02671864
Title: Impact of Incretin-mimetic Hypoglycaemic Drugs on Diabetic Retinopathy in Type 2 Diabetic Patients and Study of Biomarkers in the Development of Severe Retinopathy: Angiosafe-T2D Study 2
Brief Title: Incretin-mimetic Hypoglycemic Drugs and Severe Retinopathy
Acronym: ANGIOSAFE2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Assistance Publique Hopitaux De Marseille (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre National de la Recherche Scientifique, France (Other); Collège de France (Unknown); University of Paris 5 - Rene Descartes (Other); Pierre and Marie Curie University (Other); University Paris 7 - Denis Diderot (Other); Aix Marseille Université (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P150601
Record Dates: First submitted 2016-01-29; First posted 2016-02-02 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Type 2 Diabetes
Keywords: Incretin-based therapy; GLP1; Angiogenesis Inflammation; Hypoglycaemic treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: incretin-based therapy (Other): Patients with incretin-based therapy
  Interventions: Other: 1: incretin-based therapy
- 2: other antidiabetic (Other): Patients with other antidiabetic
  Interventions: Other: 2: other antidiabetic

INTERVENTIONS:
Other: 1: incretin-based therapy
  Arms: 1: incretin-based therapy
Other: 2: other antidiabetic
  Arms: 2: other antidiabetic

SUMMARY:
Experimental data suggest that GLP-1 promote endothelial cell growth and angiogenesis which may have beneficial effects on the cardiovascular system but harmful effects on the retina . This project investigate the possible link between incretin therapy and Severe Diabetic Retinopathy. The prevalence of severe DR in patients exposed to incretin therapy (GLP-1 analogs or DPP4 inhibitors) is compared to that in non-exposed patients to these antidiabetic classes.

DETAILED DESCRIPTION:
This study is dedicated to investigate the impact of routinely prescribed hypoglycaemic treatments on the prevalence of severe retinopathy and to seek possible biomarkers of severe retinopathy. Hypoglycemic treatments taken by the patients are those prescribe by the usuel diabetogist in the context of routine care.

The study includes T2D patients according to ADA criteria treated with any kind of hypoglycemic treatment and attending a diabetes center (three in Marseille: Department of Endocrinology, Hôpital Nord, Assistance Publique des Hôpitaux de Marseille and Service d'Ophtalmologie, Hôpital Saint-Joseph and Service de Diabétologie, Hôpital Saint-Joseph, and two in Paris : Centre Universitaire du Diabète et de ses Complications Hôpital Lariboisière, Université Paris 7, Assistance Publique des Hôpitaux de Paris and Service d'Endocrinologie, Diabétologie et Nutrition, Hôpital Bichat).

It consists of two visits: Visits1 "Inclusion" and Visits 2 "three years after the inclusion". In each visit, the investigators will collect results of eye examination (fundus) and annual diabetes check up including anthropometric data, routine biology, diabetes complication status as well as medications taken by the patients (past and current). A bio-banking (blood, urine and hairs) will be also collected. Primary objective : to compare the prevalence of severe DR in patients exposed to incretin therapy (GLP-1 analogs or DPP4 inhibitors) to that in non-exposed patients at baseline.

Secondary objective: To compare the proportion of patients who worsen DR between V1 (inclusion) and V2 (after 3-yr of treatment) in patients exposed to incretin-based therapy from baseline vs non-exposed patients: patients with no DR or mild to moderate non proliferative DR at V1 who progress to severe DR at V2.

To evaluate whether the concentrations of angiogenic/inflammatory molecules and circulating endothelial and inflammatory cells are associated with severe DR in relation with the use of GLP-1 based therapy at V1 and V2.

ELIGIBILITY:
Inclusion Criteria:

* T2D patients according to ADA criteria treated with any kind of hypoglycaemic treatment
* Age above 18 years

Exclusion Criteria:

* Type 1 diabetes
* Patients with cataract preventing DR grading
* Patients who had panretinal photocoagulation more than 10 years ago
* Documented pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7200 (Estimated)
Dates: Start 2016-04-11 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2025-04-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Severe DR at V1 (inclusion) | at inclusion
  Retinography

SECONDARY OUTCOMES:
Prevalence of severe DR at V2 (after 3 years of treatment) | after 3 years
  Retinography
Plasma concentrations of ANGPT4 | at inclusion and 3 years
Plasma concentrations of VEGF | at inclusion and 3 years
Plasma concentrations of proinflammatory cytokines such as IL-1beta, IL-6, IL-8, TNF-alpha | at inclusion and 3 years
Concentrations of blood circulating EPCs and PBMCs | at inclusion and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: GAUTIER Jean-François, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hôpital de la Conception, Marseille
  - Département de Diabétologie - Hopital Lariboisière, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaborit B, Julla JB, Besbes S, Proust M, Vincentelli C, Alos B, Ancel P, Alzaid F, Garcia R, Mailly P, Sabatier F, Righini M, Gascon P, Matonti F, Houssays M, Goumidi L, Vignaud L, Guillonneau X, Erginay A, Dupas B, Marie-Louise J, Autie M, Vidal-Trecan T, Riveline JP, Venteclef N, Massin P, Muller L, Dutour A, Gautier JF, Germain S. Glucagon-like Peptide 1 Receptor Agonists, Diabetic Retinopathy and Angiogenesis: The AngioSafe Type 2 Diabetes Study. J Clin Endocrinol Metab. 2020 Apr 1;105(4):dgz069. doi: 10.1210/clinem/dgz069. PMID 31589290